CLINICAL TRIAL: NCT02716428
Title: A Phase 2, Open-Label Study to Investigate the Safety and Efficacy of Faldaprevir and TD 6450 Alone and in Combination With Other Antivirals for 12 Weeks in Treatment-Naive Patients Chronically Infected With Genotype 1 Hepatitis C Virus
Brief Title: A Study of Faldaprevir, TD-6450 and Other Antivirals in Participants With Genotype 1b Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trek Therapeutics, PBC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRK-450-0203
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis C Viral Infection; Chronic Hepatitis C; Hepatitis C (HCV); Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — faldaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): 12 weeks of Faldaprevir plus TD-6450 plus Ribavirin
  Interventions: Drug: Faldaprevir; Drug: TD-6450; Drug: Ribavirin
- Cohort 2 (Experimental): 12 weeks of Faldaprevir plus TD-6450
  Interventions: Drug: Faldaprevir; Drug: TD-6450

INTERVENTIONS:
Drug: Faldaprevir
  Other Names: BI 201335
Drug: TD-6450
Drug: Ribavirin
  Other Names: Ribasphere®
  Arms: Cohort 1

SUMMARY:
Phase 2 study designed to assess the safety, efficacy, and pharmacokinetics of Faldaprevir and TD-6450 alone or in combination with other antivirals for a 12-week treatment duration in treatment-naïve participants with genotype 1b hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
A study to evaluate the safety and effect of treatment with experimental antiviral drugs alone or in combination with ribavirin in treatment-naïve participants with genotype 1b hepatitis C infection. The study will test the safety and anti-viral activity of two regimens administered for a duration of 12 weeks. Secondary objectives of this study are to determine the pharmacokinetics of the study drugs when co-administered, and to evaluate HCV RNA kinetics during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1b hepatitis C infection and HCV RNA ≥ 10^4 IU/mL at screening
* Hepatitis C virus treatment naive, defined as defined as having never received a direct acting anti-viral (DAA), and as having received ≤ 8 weeks of interferon ≥ 6 months prior to screening
* Absence of cirrhosis as defined by one of the following:

  * A liver biopsy performed within 24 calendar months of Day 1 showing absence of cirrhosis
  * Transient elastography (FibroScan®) performed within 12 calendar months of Day 1 with a result of ≤ 12.5 kPa (kilopascals)
  * A non-invasive test measuring liver scarring (FibroSure®) score ≤ 0.48 and AST (aspartate aminotransferase):platelet ratio (APRI) ≤ 1 performed during screening

Exclusion Criteria:

* Infection with hepatitis B virus (HBV) or human immunodeficiency virus, HIV-1 or HIV-2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving 12-week sustained virologic response following treatment with 2 direct acting anti-virals with and without ribavirin in Genotype 1b Hepatitis C infected adults | Post Treatment Week 12

SECONDARY OUTCOMES:
Percentage of subjects with virologic response 2, 4 and 8 weeks after treatment completion (HCV RNA less than lower limit of quantitation at 2, 4 and 8 weeks after end of therapy with Faldaprevir plus TD-6450 with and without ribavirin) | Post Treatment Weeks 2 to 8
Safety as determined by the incidence of serious adverse events, Grade 3 or 4 adverse events and laboratory abnormalities, and discontinuations due to adverse events | Randomization through End of Study, up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ed Gane, MD, Principal Investigator — Auckland Clinical Studies Ltd; Tarek Hassanein, MD, Principal Investigator — Southern California Research Center
Locations (6):
- United States (3):
  - Southern California Research Center, Coronado, California
  - Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - Gastro One, Germantown, Tennessee
- New Zealand (3):
  - Auckland Clinical Studies, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Waikato

IPD SHARING:
Plan to Share IPD: No